CLINICAL TRIAL: NCT06995300
Title: Minimally Invasive Isolated Decompression From the Posterior Approach for Degenerative Spinal Stenosis of the Cervical Spine
Brief Title: Minimally Invasive Posterior Decompression of the Cervical Spine
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: N.N. Priorov National Medical Research Center of Traumatology and Orthopedics (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NS12-03
Record Dates: First submitted 2025-05-12; First posted 2025-05-29 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-05

CONDITIONS: Cervical Degenerative Disc Disease; Cervical Stenosis; Posterior Spine Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohort (Other): All patients will undergo minimally invasive isolated decompression via the posterior approach to the cervical spine
  Interventions: Procedure: minimally invasive decompression via the posterior approach

INTERVENTIONS:
Procedure: minimally invasive decompression via the posterior approach — All patients will undergo minimally invasive isolated decompression via the posterior approach to the cervical spine.

SUMMARY:
Degenerative stenosis of the cervical spinal canal may be caused by the compression of the posterior part of the dural sac and spinal cord by the hypertrophied ligamentum flavum and facet joints, by the compression of the anterior part of the dural sac and spinal cord by the posterior longitudinal ligament, vertebral osteophytes and protrusion/ herniation.

The choice of surgical treatment in such cases is challenging. Posterior decompression and fixation is often proposed, but it is associated with a traumatic posterior approach, a large wound, and blood loss, a high risk of surgery site infections, and also instability of the metal fixation is possible. Also important is the increase in the surgical procedure cost due to the use of metal implants. An excellent alternative to standard posterior decompression and fixation is a method with isolated decompression of the cervical canal via posterior approach, which does not require any metal fixation.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years old;
2. Degenerative symptomatic cervical stenosis caused by posterior compression (hypertrophied ligament flavum and/or hypertrophied facet joints etc.) confirmed by MRI;
3. Symptoms persisting for at least 3 months prior to surgery;
4. Planned surgical decompression for one and more cervical level;
5. Given written Informed Consent;
6. Able and agree to fully comply with the clinical protocol and willing to adhere to follow-up schedule and requirements.

Exclusion Criteria:

1. The need for anterior cervical decompression;
2. Prior cervical fusion at any level;
3. Any contraindication or inability to undergo baseline and/or follow up MRI or X-ray as required per protocol;
4. Neck or non-radicular pain of unknown etiology;
5. History or presence of any other major neurological disease or condition that may interfere with the study assessments;
6. Previous enrollment in this study, current enrollment or plans to be enrolled in another study (in parallel to this study).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2026-05-19 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change in the cross-sectional area of the dural sac, mm2 | 3 months after surgery
  To observe the change in the cross-sectional area of the dural sac by MRI

SECONDARY OUTCOMES:
Change from baseline in Japanese Orthopaedic Association scale | 3 months and 12 months postoperatively
  To observe the change from baseline in Japanese Orthopaedic Association scale at 3 months after surgery (0 points - the severest myelopathy, 17 points - no myelopathy)
Change from baseline in Neck Disability Index | 2 weeks (or at day of hospital discharge), 3 months, 12 and 12 months postoperatively
  To observe the change of Oswestry Disability Index as compared to baseline through follow-up terms (min - 0 - the best result, patient is active; max - 50 - the worst result, patient is not physically active)
Change from baseline in The Health Transition Item from SF-36 | 2 weeks (or at day of hospital discharge), 3 months, 12 months postoperatively
  To observe the change of The Health Transition Item as compared to baseline through follow-up terms (Patient's answers range from ''Much Better,'' ''Somewhat Better,'' ''About the Same,'' ''Somewhat Worse,'' to ''Much Worse.'')
Change in the cross-sectional area of the dural sac, mm2 | 12 months postoperatively
  To observe the change in the cross-sectional area of the dural sac by MRI
Change from baseline in cervical balance parameters | 3 months and 12 months postoperatively
  To observe the change of regional balance parameters - Cervical Lordosis - by sagittal scans of cervical spine by X-Ray compared to baseline, in degrees
Change from baseline in cervical balance parameters | 3 months and 12 months postoperatively
  To observe the change of regional balance parameters - Segmental Lordosis - by sagittal scans of cervical spine by X-Ray compared to baseline, in degrees
Change from baseline in cervical balance parameters | 3 months and 12 months postoperatively
  To observe the change of regional balance parameters - C2-C7 Sagittal Vertical Axis - - by sagittal scans of cervical spine by X-Ray compared to baseline, in degrees
Adverse Events | during study, an average of 1 year
  Document Adverse Events (incl. adverse events related to device) occurrence throughout the study
Change from baseline in Numeric Pain Rating Scale | 2 weeks (or at day of hospital discharge), 3 months, 12 months postoperatively
  To observe the change of Numeric Pain Rating Scale as compared to baseline through follow-up terms (0 - no pain, 10 - unbearable pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Priorov National Medical Research Center of Traumatology and Orthopedics, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No